CLINICAL TRIAL: NCT07245927
Title: An Open, Prospective, Non-interventional, Multicentre, Controlled Study of Safety and Efficacy of the Thrombolysis With the Non-immunogenic Staphylokinase in Patients With Massive Pulmonary Embolism (FORPE Registry)
Brief Title: Post-registration Trial of the Non-immunogenic Staphylokinase in Massive Pulmonary Embolism
Status: Recruiting | Type: Observational
Sponsor: Supergene, LLC (Industry)
Collaborators: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Other Study IDs: FORPE Registry
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Embolism Acute Massive
Keywords: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-immunogenic staphylokinase: Drug: non-immunogenic staphylokinase 15 mg as a single intravenous bolus Other Names: Fortelyzin®
  Interventions: Drug: Non-immunogenic staphylokinasenon-immunogenic staphylokinase 15 mg as a single intravenous bolus Other Names: Fortelyzin®

INTERVENTIONS:
Drug: Non-immunogenic staphylokinasenon-immunogenic staphylokinase 15 mg as a single intravenous bolus Other Names: Fortelyzin® — Non-immunogenic staphylokinase 15 mg as a single intravenous bolus
  Other Names: Fortelyzin®

SUMMARY:
The aim of FORPE Registry is to study the safety and efficacy of the non-immunogenic staphylokinase in patients with massive pulmonary embolism in routine clinical practice.

DETAILED DESCRIPTION:
In November 2023 a multicenter, open-label, randomized non-inferiority trial of the efficacy and safety of the non-immunogenic staphylokinase (Fortelyzin®) compared with alteplase (Actilyse®) in patients with massive pulmonary embolism (FORPE) has been completed (NCT04688320).

FORPE trial is the first report of the non-immunogenic staphylokinase usage in patients with massive pulmonary embolism accompanied by unstable haemodynamics. Non-immunogenic staphylokinase was found to be non-inferior to alteplase (p=1.00). Non-immunogenic staphylokinase had high safety profile and did not cause the major bleeding. No cases of haemorrhagic stroke or major bleeding were recorded in the non-immunogenic staphylokinase group, whereas there were five cases (5%) of BARC type 3+5 bleedings in the alteplase group (p=0.026). All major bleedings and fatal intracranial haemorrhage in the alteplase group were registered only in 60 years old patients.

The unique mechanism of action of non-immunogenic staphylokinase allows it to be used in a single dose of 15 mg, regardless of the patient's body weight. Non-immunogenic staphylokinase is easy to administer with a rapid single bolus that makes it convenient for use in emergency medicine.

The indication "massive pulmonary embolism" is included in the Instructions for medical use of the non-immunogenic staphylokinase. In routine clinical practice, the non-immunogenic staphylokinase is used for massive pulmonary embolism treatment since 2024.

The aim of FORPE Registry is to study the safety and efficacy of the non-immunogenic staphylokinase in patients with massive pulmonary embolism in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and older.
* Verified diagnosis of massive pulmonary embolism (using computer tomography)
* Signs of overload / dysfunction of the right ventricle (at least one) in combination with persistent arterial hypotension or shock
* The time from the symptoms onset is no more than 14 days.
* Thrombolysis with the non-immunogenic staphylokinase, 15 mg as a single intravenous bolus.

Exclusion Criteria:

* Increased risk of bleeding:

  * extensive bleeding at present or within the previous 6 months;
  * intracranial (including subarachnoid) hemorrhage at present or in history;
  * hemorrhagic stroke within the last 6 months;
  * a history of diseases of the central nervous system (including neoplasms, aneurysms);
  * intracranial or spinal surgical interventions within the last 2 months;
  * major surgery or major trauma within the previous 4 weeks;
  * recent puncture of an incompressible blood vessel (eg, subclavian or jugular vein);
  * severe liver disease, including liver failure, cirrhosis, portal hypertension (including esophageal varices) and active hepatitis;
  * confirmed gastric or duodenal ulcer within the last 3 months;
  * neoplasm with an increased risk of bleeding;
  * simultaneous administration of Dabigatran without prior administration of idarucizumab;
  * arterial aneurysms, developmental defects of arteries / veins;
  * acute pancreatitis;
  * bacterial endocarditis, pericarditis;
  * suspicion of aortic dissecting aneurysm;
  * any other conditions, in the opinion of the investigator, associated with a high risk of bleeding.
* Lactation, pregnancy.
* Known hypersensitivity to the non-immunogenic recombinant staphylokinase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 18 years and older with verified massive pulmonary embolism, who received a single intravenous bolus of the non-immunogenic staphylokinase (15 mg).
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | day 7 after drug administration
  The number of death from any causes during admission

SECONDARY OUTCOMES:
All-cause mortality | day 30 after drug administration
  The number of death from any causes during 30 days after drug administration
Haemodynamic Collapse | day 30 after drug administration
  The number of haemodynamic collapses from any causes during 30 days after drug administration
Recurrent Pulmonary Embolism | day 30 after drug administration
  The number of recurrent pulmonary embolism from any causes during 30 days after drug administration
Pulmonary Artery Systolic Pressure Measures | baseline and day 2 after drug administration
  The efficacy is evaluated in terms of pulmonary artery systolic pressure after drug administration

OTHER OUTCOMES:
Intracranial haemorrhage | day 30 after drug administration
  The number of intracranial haemorrhage during 30 days after drug administration
Major bleedings | day 30 after drug administration
  The number of major bleedings (according to BARC classification type 3 and 5) during 30 days after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Sergei S. Markin, MD, Prof., Study Director — LLC "SuperGene"
Locations (1):
- E.I. Chazov National Medical Research Center of Cardiology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kirienko AI, Leontyev SG, Tereschenko SN, Yavelov IS, Shakhnovich RM, Erlikh AD, Talibov OB, Yarovaya EB, Semenov AM, Semenov MP, Ivanov SV, Beregovykh VV, Archakov AI, Markin SS; FORPE study group. Non-immunogenic recombinant staphylokinase versus alteplase for patients with massive pulmonary embolism: a randomized open-label, multicenter, parallel-group, non-inferiority trial, FORPE. J Thromb Haemost. 2025 Feb;23(2):657-667. doi: 10.1016/j.jtha.2024.09.035. Epub 2024 Oct 23. PMID 39454884
- [Result] Leontyev SG, Yarovaya EB, Kutsenko VA, Ivlev OE, Soplenkova AG, Semenov AM, Semenov MP, Ivanov SV, Romashova YA, Markin SS. The Safety of Non-immunogenic Recombinant Staphylokinase in Elderly Patients With Massive Pulmonary Embolism: A Randomized Clinical Trial FORPE. Health Sci Rep. 2025 May 19;8(5):e70826. doi: 10.1002/hsr2.70826. eCollection 2025 May. PMID 40391253